CLINICAL TRIAL: NCT03390660
Title: Trends in Breastfeeding Disparity in U.S. Infants by WIC Eligibility and Participation: Evidence From NHANES 1999-2014
Brief Title: Trends in Breastfeeding Disparity in U.S. Infants by WIC Eligibility and Participation
Acronym: WIC breastfeed
Status: Completed | Type: Observational
Sponsor: Old Dominion University (Other)
Responsible Party: Principal Investigator, Qi Zhang, Associate Professor, Old Dominion University
Other Study IDs: 2017-001
Record Dates: First submitted 2017-12-28; First posted 2018-01-04 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2017-12

CONDITIONS: Breast Feeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- birth cohorts: born in 1994-1997, 1998-2001, 2002-2005, 2006-2009, 2010-2014
  Interventions: Other: WIC program participation

INTERVENTIONS:
Other: WIC program participation — WIC program is a welfare program in the U.S. to provide nutritional supplements to low-income women, infants, and children.

SUMMARY:
This is a secondary data analysis study that uses nationally representative data to examine the trends in breastfeeding disparities between Women, Infants, and Children (WIC) program eligible children vs. non-eligible children and eligible participants vs. eligible non-participants.

ELIGIBILITY:
Inclusion Criteria:

* infants or children surveyed in NHANES 1999-2014 aged younger than 72 months

Exclusion Criteria:

* infants or children with missing information in breastfeeding, WIC participation, or other major socio-demographics, such as income

Ages: 1 Month to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A nationally representative sample surveyed in NHANES 1999-2014
Sampling Method: Probability Sample
Enrollment: 13771 (Actual)
Dates: Start 1999-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Everbreastfeeding | till age 5
  whether the child has ever been breastfed
Breastfeeding at 6 months | till age 6 months
  whether the child was breastfed at age 6 months

IPD SHARING:
Plan to Share IPD: No